CLINICAL TRIAL: NCT00453258
Title: Analysis of Human Tear Proteins: A Pilot Study to Describe the Tear Film Proteome of Patients Undergoing Ophthalmic Examination.
Brief Title: Pilot Study of Human Tear Proteins
Status: Terminated | Type: Observational
Why Stopped: Stopped due to low enrollment
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0862
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2012-10

CONDITIONS: Eye Disease
Keywords: ocular proteomics; eye disease; proteomics
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Subject: Subjects receiving eye examination
  Interventions: Other: Eye Examination

INTERVENTIONS:
Other: Eye Examination — Subjects receiving eye examination

SUMMARY:
The significance of our study is in the importance of understanding the quality and quantity of proteins in the human tear film from diseased and non-diseased patients. This pilot study will provide data to plan prospective research to better delineate the utility of tear proteins in diagnosing and following disease status in a non-invasive fashion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* able to cooperate with tear sample collection
* provide written informed consent

Exclusion Criteria:

* special populations (children, pregnant or lactating females, prisoners, etc)
* refusal to sign sudy consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects receiving eye examination
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2007-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plan Prospective Research | Throughout study participation
  Pilot study will provide data to plan prospective research to better delineate the utility of tear proteins in diagnosing and following disease status in a non-invasive fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Malik Y. Kahook, MD, Principal Investigator — Rocky Mountain Lions Eye Institute
Locations (1):
- Rocky Mountain Lions Eye Institute, Aurora, Colorado, United States